CLINICAL TRIAL: NCT05551585
Title: A Randomized, Double-blind, Sham-controlled Clinical Trial of Transcranial Pulse Stimulation for the Treatment of Major Depression
Brief Title: Transcranial Pulse Stimulation for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSEARS20220816001-02
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Major Depression
Keywords: Transcranial pulse stimulation; Brain stimulation; Major depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real TPS treatment group (Experimental): 1. Participants with MDD will receive TPS treatment lasting for 4 weeks (3 sessions per week).
  2. A follow-up assessment will be scheduled 3 months after the last REAL treatment day.
  3. MRI measurements will be conducted before the start of treatment (within one week before treatment start), as well as after the last treatment day (within one week post-treatment)
  Interventions: Device: Transcranial pulse stimulation
- Sham TPS treatment (Sham Comparator): 1. Participants will receive sham TPS treatment lasting for 4 weeks (3 sessions per week, as done previously.
  2. After treatment end and completed assessments, the study will be unblinded and participants in the sham treatment arm will receive real TPS.
  3. A follow-up assessment will be scheduled 3 months after the last REAL treatment day.
  4. MRI measurements will be conducted before the start of treatment (within one week before treatment start), as well as after the last treatment day (within one week post-treatment),
  Interventions: Device: Transcranial pulse stimulation

INTERVENTIONS:
Device: Transcranial pulse stimulation — TPS will be performed in three treatment sessions per week, applying 1000 pulses per session (single ultrashort (3 μs) ultrasound pulses, 0.2-0.25 mJ mm-2, ~5 Hz pulse frequency,

SUMMARY:
Transcranial pulse stimulation (TPS) is a newly developed brain stimulation therapy from Austria & Germany with highly promising applicability in neuropsychiatric disorders. Major depressive disorder (MDD) is the world's leading cause of disability. Novel treatment approaches are urgently needed given that a significant fraction of patients does not sufficiently respond to standard antidepressant treatments. Our open-label pilot study using TPS in MDD indicates preliminary efficacy. However, experimental control is necessary to infer reliable scientific evidence for the efficacy of TPS. Here, we propose a randomized, double-blind, sham-controlled clinical trial to probe the utility of TPS as a modern antidepressant treatment.

ELIGIBILITY:
MDD group

Inclusion Criteria:

* Age 18 to 65;
* A clinical diagnosis of a MDD according to psychiatrist visit records or a clinical interview using the Chinese version of the Mini International Neuropsychiatric Interview (MINI)
* Baseline HAMD17 score ≥ 14;
* Treatment naivety or stable (≥4 weeks) psychopharmacological medication.

Exclusion Criteria:

* Severe internal diseases including blood clotting disorders;
* Neurological disorders including bleeding prone micro-pathologies or a history of severe head injuries;
* Current psychiatric comorbidities, including addiction;
* Pregnancy;
* Common NIBS exclusion criteria, such as a history of brain surgery, cardiac pacemaker, deep brain stimulation and intracranial metallic particles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms after the treatment | four weeks of treatment
  Primary clinical outcome measure will be a change in Montgomery-Åsberg Depression Rating Scale (MADRS) score (range from 0-60) after six weeks of treatment. Higher scores indicative of greater depressive symptomology in MADRS

SECONDARY OUTCOMES:
Change in depressive symptoms in the follow-up stage | at 3 months follow-up
  Change of Montgomery-Åsberg Depression Rating Scale (MADRS) score (range from 0-60) at 3-months follow-up. Higher scores indicative of greater depressive symptomology in MADRS.
Change in depressive symptoms | four weeks of treatment and at 3 months follow-up
  Change of Hamilton Depression Rating Scale (HAMD17, range from 0-54) scores after four weeks of treatment and at 3-months follow-up. Higher scores indicative of greater depressive symptomology in HAMD-17
Change in depressive symptoms | four weeks of treatment and at 3 months follow-up.
  Change of Patient Health Questionnaire (PHQ-9, range from 0-27) scores after four weeks of treatment and at 3-months follow-up. Higher scores indicative of greater depressive symptomology in PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Georg S. Kranz, PhD, Principal Investigator — The Kong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No